CLINICAL TRIAL: NCT00417690
Title: A Prospective Randomized Double-Blind Study of PASER® in the Management of Patients Experiencing an Acute Flare of Crohn's Disease
Brief Title: High Dose Oral 4-Aminosalicylic Acid (PASER®) to Control Acute Flares of Mild to Moderate Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efforts at recruitment have halted as recruitment was poor.
Sponsor: Jacobus Pharmaceutical (Industry)
Responsible Party: Kathy Ales, MD Medical Director, Jacobus Pharmaceutical Company, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PASER-AFC.001
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Crohn's Disease
Keywords: Crohn's Disease; Acute Flare; Mild to moderate Crohn's Disease; Ileocecal distribution
MeSH Terms: conditions — Crohn Disease | interventions — Aminosalicylic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental): Oral granules administered as one 4 g packet three times daily for two weeks followed by one 4 g packet two times daily for two weeks
  Interventions: Drug: 4-Aminosalicylic acid
- P (Placebo Comparator): One packet of oral granules administered three times daily for 2 weeks followed by one packet two times daily for two weeks
  Interventions: Drug: PASER placebo granules

INTERVENTIONS:
Drug: 4-Aminosalicylic acid — Oral granules administered as one 4 g packet three times daily for two weeks followed by one 4 g packet two times daily for two weeks
  Other Names: PASER Granules; NDC 49938-107-04
  Arms: A
Drug: PASER placebo granules — Oral granules administered administered as one packet three times daily for two weeks followed by one packet two times daily for two weeks
  Arms: P

SUMMARY:
The purpose of this 4 week study is to determine whether PASER®, an approved delayed-release oral formulation of 4-aminosalicylic acid, in doses of 4 grams three times daily for 2 weeks followed by 4 grams twice daily for 2 weeks, will resolve an acute flare of ileocecal Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Crohn's disease involving predominantly the ileum and/or cecum. The diagnosis must have been established by radiography, endoscopy and/or biopsy (at least 2 of the 3 modalities) with at least one confirmatory test having been performed no more than 36 months before entry. The diagnosis must have been confirmed by at least one gastroenterologist.
* Harvey Bradshaw Index of at least 7
* The onset of the acute flare should have been abrupt, declaring itself over 72 hours, and should have started no more than 4 weeks before study entry. Symptoms relating to the flare should not have diminished or started to improve prior to entry.
* Written informed consent

Exclusion Criteria:

* Concomitant corticosteroids, including budesonide
* Corticosteroids within the previous 2 months
* Cyclosporine, mycophenolate mofetil or experimental drugs during the last three months
* Maintenance infliximab, or infliximab or other biologics in the preceding 3 months
* Change in dose during previous 4 weeks in 5-aminosalicylate, probiotic and/or antibiotic, or in chronic azathioprine, 6-mercaptopurine, or methotrexate
* If currently using azathioprine, 6-mercaptopurine or methotrexate, these must have been used steadily for at least 4 months
* Current experimental drugs or experimental drugs within the last 3 months
* If the severity of the flare has started to decrease spontaneously
* Coexisting diagnosis of primary sclerosing cholangitis,
* Infectious diarrhea,
* Signs of intestinal obstruction or perforation or abscess,
* New fistulization as part of the acute flare or increased activity in chronic fistula(e) as part of the acute flare,
* Increased activity of pre-existing anal or rectal Crohn's disease as part of the flare
* Allergy or sensitivity to salicylates
* Pregnancy or breast-feeding
* Failure of a woman of child-bearing age to agree to use adequate contraception for the 4 week period of the trial, if sexually active
* Severe renal or hepatic disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Response, as defined by a reduction of the CDAI score of >70 points by 4 weeks compared with baseline | 4 weeks

SECONDARY OUTCOMES:
Rate of remission as defined by the decrease in CDAI > 100 points and total CDAI < 150 by 4 weeks | 4 weeks
Rate of response as defined by a reduction in HBI to less than 5 by 4 weeks | 4 weeks
Rate of remission as defined by the decrease in HBI to less than 3 by 4 weeks | 4 weeks
Time to response and/or remission including time to change in HBI, according to elements of the daily patient diary | up to 4 weeks
Increase in IBDQ to greater than 170 and the time to score above 170 | 4 weeks
The change from baseline in the patient's general sense of disease activity as recorded in the individual daily diary | up to 4 weeks
Absence of night time stools, if they were present on entry, and time to disappearance | up to 4 weeks
Time to normalization of all other components in the diary | up to 4 weeks
Change in Hgb, ESR, CRP, platelet count, calprotectin from baseline and time to normalization | 2 weeks and 4 weeks
Change in global physician assessment of disease activity from baseline to study completion | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David P. Jacobus, MD, Study Chair — Jacobus Pharmaceutical; Kathy L. Ales, MD, Study Director — Jacobus Pharmaceutical; Daniel Present, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Stephen B. Hanauer, MD, Principal Investigator — University of Chicago Hospitals; John Hanson, MD, Principal Investigator — Charlotte Gastroenterology & Hepatology, PLLC; Iris Dotan, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center; Rami Eliakim, MD, Principal Investigator — Rambam Health Care Campus
Locations (5):
- United States (3):
  - The University of Chicago, Chicago, Illinois
  - Mount Sinai School of Medicine IBD Research Center, New York, New York
  - Charlotte Gastroenterology and Hepatology, PLLC, Charlotte, North Carolina
- Israel (2):
  - Rambam Medical Center, Haifa
  - Tel-Aviv Sourasky Medical Center, Tel Aviv